CLINICAL TRIAL: NCT00752635
Title: Comparison of Efficacy and Safety of Tricilest (Norgestimate-ethinyl Estradiol) and Diane-35 (Cyproterone Acetate-ethinyl Estradiol) in the Treatment of Acne Vulgaris
Brief Title: Comparison of Efficacy and Safety of Norgestimate-ethinyl Estradiol and Cyproterone Acetate-ethinyl Estradiol in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Taiwan Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR007129
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Acne Vulgaris
Keywords: TriCilest; acne vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Moxifloxacin; Cyproterone acetate, ethinyl estradiol drug combination

INTERVENTIONS:
Drug: Norgestimate-ethinyl estradiol; Cyproterone acetate-ethinyl estradiol

SUMMARY:
The purpose of this study was to evaluate the effectiveness and safety of norgestimate-ethinyl estradiol as comparted with cyproterone acetate-ethinyl estradiol among female patients with moderate acne vulgaris.

DETAILED DESCRIPTION:
This study was to evaluate the efficacy and safety of TriCilest as comparted with Diane-35 among female patients with moderate acne vulgaris. The study design was double-blind, randomized, parallel and active controlled. The sponsor planned to recruit approximately 50 patients to complete 40 evaluable patients. At the end of the study, a total of 48 patients were randomized.

TriCilest (noregestimate-ethinyl estradiol), 0.18mg-0.035mg or 0.215mg-0.035mg or 0.25mg-0.035mg, Oral admistration, The duration was three consecutive menstrual cycles.

ELIGIBILITY:
Inclusion Criteria:

* Female adults who were suffering from moderate acne vulgaris (grade II or III)
* With 6 to 100 comedones (non-inflammatory lesions)
* With 10 to 50 inflammatory lesions (papules or pustules)
* With fewer than 5 nodules
* Agree to condoms or diaphragm, and spermicide or any other medically approved effective barrier method of contraceptive or a nonhormonal IUD
* Agree to take as treatment for acne only for the supplied study drug during the three month treatment phase
* Documented by an informed consent to participate in the trial on the day before entering the study

Exclusion Criteria:

* Patients who, in the investigator's opinion, cannot understand or follow the instructions given in the study
* Who are pregnant or nursing
* Who have clinical depression and are suicidal or require immediate treatment for depression
* Who have a known hypersensitivity to any of the ingredients
* Who are currently having significant adverse experiences from ethinyl estradiol or norgestimate
* Who have any coexisting medical condition or are taking and concomitant to a medication that is likely to interfere with safe administration of TriCilest and/or Diane-35, in the investigator's opinion
* Who take systemic retinoids, systemic antimicrobials, and topical acne treatments within 6 months, 1 month, and 2 weeks prior to enrollment, respectively
* Who have any of the following contraindications to oral contraceptives: Current thrombophlebitis or thromboembolic disorders, or past history of deep vein thrombophlebitis or thromboembolic disorder, or cerebral vascular or coronary artery disease or known severe hypertension, or diabetes with vascular involvement, or known or suspected carcinoma of the breast, or known or suspected estrogen-dependent neoplasia, or undiagnosed, abnormal genital bleeding, or benign or malignant liver tumor, or have jaundice or severe liver disease, or neurovascular lesion of the eye or serious visual disturbances, or known allergic reaction or sensitivities to TriCilest or Diane 35
* Who have taken an investigational medication within 30 days prior to enter study (or within a period of five times its half-life or the half-life of its metabolites)

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2004-09; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable was the change form baseline to the latest available evaluation in total lesion count. The primary efficacy result of this study clearly manifested the potency of TriCilest.

SECONDARY OUTCOMES:
The secondary efficacy variable (change in lesion counts) showed consistent results to the primary efficacy endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Taiwan, Ltd. Clinical Trial, Study Director — Johnson & Johnson Taiwan Ltd

REFERENCES:
- See also: Comparison of efficacy and safety of Tricilest (norgestimate-ethinyl estradiol) and Diane-35 (cyproterone acetate-ethinyl estradiol) in the treatment of acne vulgaris — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=693&filename=CR007129_CSR.pdf